CLINICAL TRIAL: NCT04139486
Title: adaptatiVe Endovascular Strategy to the CloT MRI in Large Intracranial Vessel Occlusion
Acronym: VECTOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Collaborators: University Hospital, Lille (Other); Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC19_0174
Record Dates: First submitted 2019-10-07; First posted 2019-10-25 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: Intracranial Thrombosis
Keywords: Contact aspiration (CA); Embotrap II; Susceptibility vessel sign (SVS); Thrombus; Embotrap III
MeSH Terms: conditions — Intracranial Thrombosis; Thrombosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Open-label study with blinded evaluation (PROBE)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combined EMBOTRAP II or III and Contact Aspiration (Experimental)
  Interventions: Procedure: combined EMBOTRAP II or III and Contact Aspiration
- Contact Aspiration alone (Active Comparator)
  Interventions: Procedure: Contact Aspiration alone

INTERVENTIONS:
Procedure: combined EMBOTRAP II or III and Contact Aspiration — refer to title
  Arms: combined EMBOTRAP II or III and Contact Aspiration
Procedure: Contact Aspiration alone — refer to title
  Arms: Contact Aspiration alone

SUMMARY:
In the VECTOR trial, the aim is to analyze, in case of SVS+ occlusions, a first line Embotrap II added to CA combined strategy compare to CA alone strategy.

Many practitioners are convinced that a first line strategy with CA alone is easy, safe, rapid and efficient. Maybe, after two, three, four ... passes and with the secondary help of a combined strategy, a high rate of eTICI 2b/3 could be reached with a CA first line strategy. But this could go with a higher number of passes, a waste of time and a suboptimal angiographic results (eTICI 2b) due to distal emboli, especially in case of friable, non-well organized, red blood cell rich (RBC) i.e. SVS + thrombi (25-28). This could, be related to worst clinical outcome at 3 months. VECTOR asks a relevant question: Do the invetigators have to add the use of an Embotrap II or III to the CA, from the first passes, in case of SVS+ clots?

DETAILED DESCRIPTION:
Sudden occlusion of an intracranial artery by a thrombus represents the initial and pivotal event of large vessel occlusion acute ischemic stroke (AIS). The primary goal of AIS treatment is to re-open this artery with intravenous tissue-type plasminogen activator infusion (IV t-PA) and/or endovascular therapy (EVT). Thrombus characterization could be useful to predict AIS etiology, IV t-PA response and to adapt the device or technique for EVT. Especially, approaching the red blood cell (RBC) content of the thrombus would be helpful to plan a treatment strategy or identify specific EVT approaches in order to maximize the rate of early successful reperfusion .

The susceptibility vessel sign (SVS) on T2*-MRI sequence is defined as a hypo-intense signal exceeding the diameter of the contralateral artery located at the site of the thrombus. Several studies have demonstrated SVS to be a negative predictor of early reperfusion after IV t-PA and an incentive to EVT . Two studies identified a correlation between the SVS and the thrombus composition (specifically the RBC composition). In the ASTER trial, the presence of SVS impacted the success rate of the EVT strategy. In the SVS (+) sub-population of this study, compared to contact aspiration (CA), patients treated with stent retrievers achieved higher rates of complete reperfusion within fewer passes, which translated into a better functional outcome. In the absence of SVS, no differences were observed between the two techniques. Furthermore; based on the ASTER and THRACE trial populations treated with stent retriever as a first line strategy, a higher rate of favorable clinical outcome at 3 months in SVS (+) patients was recently found . Hence, that differences in terms of reperfusion results are thought to be related to different clot compositions between SVS + and SVS - occlusions.

In the VECTOR trial, the aim is to analyze, in case of SVS+ occlusions, a first line Embotrap II added to CA combined strategy compare to CA alone strategy.

Many practitioners are convinced that a first line strategy with CA alone is easy, safe, rapid and efficient. Maybe, after two, three, four passes and with the secondary help of a combined strategy, a high rate of eTICI 2b/3 could be reached with a CA first line strategy. But this could go with a higher number of passes, a waste of time and a suboptimal angiographic results (eTICI 2b) due to distal emboli, especially in case of friable, non-well organized, red blood cell rich (RBC) i.e. SVS + thrombi. This could, be related to worst clinical outcome at 3 months.

VECTOR asks a relevant question: Do the investigators have to add the use of an Embotrap II or III to the CA, from the first passes, in case of SVS+ clots? The hypothesis in the VECTOR trial is that the Embotrap II or III, thanks to its dedicated design will help to the stabilization of friable clots and allow better retrieving of SVS + thrombi in a lower number of passes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older (i.e., candidates must have had their 18th birthday)
* Puncture carried out within 24 hours of first symptoms
* Suitable 1.5T MRI T2 * Gradient echo that shows a clear susceptibility vessel sign facing the occlusion
* Neuroimaging demonstrates large vessel proximal occlusion (distal ICA through MCA bifurcation, M1 or proximal M2)
* Patient or trustworthy person informed about the study and having orally consented to participation in the study. If the patient is unable to receive information and no trustworthy person can be contacted during screening for the study, trial inclusion will be completed as an emergency procedure by the investigator, in compliance with the French laws
* With or without intravenous thrombolysis

Exclusion Criteria:

* Absence of large vessel occlusion on non-invasive imaging
* Known or suspected pre-existing (chronic) large vessel occlusion in the symptomatic territory
* Suspected pregnancy; if, in a woman is of child-bearing potential, a urine or serum beta HCG test is positive
* Severe contrast medium allergy or absolute contraindication to use of iodinated products
* Clinical history, past imaging or clinical judgment suggests that the intracranial occlusion is chronic
* Patient has severe or fatal comorbidities that will likely prevent improvement or follow-up or that will render the procedure unlikely to benefit the patient
* Acute ischemic stroke involving posterior circulation (vertebro-basilar occlusion)
* Angiographic evidence of carotid dissection or tandem cervical occlusion or stenosis requiring treatment
* Pregnant or breast-feeding women
* Patient benefiting from a legal protection
* Non-membership of a national insurance scheme
* Opposition of the patient or (in case of inclusion as a matter of urgency) of the trustworthy person
* Patient with modified Rankin score > 3 before qualifying stroke

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 526 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2022-02-14 (Actual); Study Completion 2022-10-03 (Actual)

PRIMARY OUTCOMES:
The rate of near to complete reperfusion after 3 passes of the device defined by a modified treatment in cerebral infarction (eTICI) score of 2c/3 | At Day 0 immediately after 3 passes
  Preliminary data suggested in case of SVS+ occlusions a superiority of the first line SR strategy in terms of eTICI2c/3 after 3 passes compared to first line CA alone.The first pass (FPE) is an ambitious technical endpoint defined as a successful reperfusion obtained after the first pass that has been recently associated with an increased probability of favorable clinical outcome, a reduced mortality rate and procedural adverse events.However, this constitutes a "very technical" endpoint and the external validity in daily practice would be reduced compared to the three passes cut-off.Even if a FPE eTICI 2b, 2c or 3 has shown better clinical outcome compared to a final eTICI 2b, 2c or 3,there is no study that has proved the better clinical outcome when compared FPE eTICI 2b,2c or 3 to three passes eTICI 2b,2c or 3.Last, there was no preliminary data that suggests in case of SVS+ occlusions, a superiority of the first pass SR strategy in terms eTICI2c/3 compared to first pass CA alone.

SECONDARY OUTCOMES:
Near to complete first-pass effect | Day 0 immediately after first pass
  Defined as a eTICI 2c/3 after first pass device
Complete first-pass effect | Day 0 immediately after first pass
  Defined as a eTICI 3 after first pass device
Complete reperfusion | Day 0 immediately after three passes
  Defined as eTICI 3 after three passes
Final near to complete reperfusion | Day 0 at the end of the intervention
  Defined as eTICI 2c/3 final
Final complete reperfusion | Day 0 at the end of the intervention
  Defined as eTICI 3
Time to achieve eTICI 2c or better revascularization | Day 0
  Time to achieve eTICI 2c or better revascularization
Time between groin puncture to clot contact | Day 0
  Time between groin puncture to clot contact
Rate of functional independence | At 90days
  Defined as a modified Rankin scale (mRS) 0-2
Rate of excellent functional outcome | At 90days
  Defined as a mRS 0-1
The distribution of mRs scores | At 90days
  Combining scores of 9 and 10
Change in NIHSS from baseline to 24 hours | Baseline and 24hours
  Change in NIHSS
Rate of symptomatic and asymptomatic intracerebral hemorrhage | At 24hrs
  Assessment of symptomatic and asymptomatic intracerebral hemorrhage at MRI or CT scan 24h after thrombectomy
Rate of parenchymal hematoma type 1 and 2 | At 24hrs
  Assessment of parenchymal hematoma type 1 and 2
Rate of all-cause mortality at 90 days | At 90days
  Assessment of all-cause mortality at 90 days
Rate of periprocedural complications | At 90days
  Occurrence of emboli to new territory, vasospasm, dissection, perforation and subarachnoid hemorrhage

CONTACTS AND LOCATIONS:
Overall Officials: Romain Bourcier, Principal Investigator — Nantes University Hospital
Locations (23):
- France (23):
  - CHU Amiens-Picardie, Amiens
  - CH Angers, Angers
  - CH Côte Basque, Bayonne
  - Hôpital Pellegrin - CHU Bordeaux, Bordeaux
  - CHRU Brest, Brest
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hôpital Roger Salengro - CHR Lille, Lille
  - CHU Limoges, Limoges
  - Hospices Civils Lyon, Lyon
  - CHU Marseille - Hôpital la Timone, Marseille
  - CHU Gui de Chauliac, Montpellier
  - CHU Nancy, Nancy
  - CHU de Nantes, Nantes
  - Fondation Ophtalmologique Adolphe de Rothschild, Paris
  - Hôpital Ste Anne, Paris
  - La Pitié Salpétrière, Paris
  - CH PAU, Pau
  - Hôpital Maison Blanche - CHU Reims, Reims
  - Hôpital Pontchaillou - CHU Rennes, Rennes
  - CHU Strasbourg, Strasbourg
  - Hôpital FOCH, Suresnes
  - Hôpital Bretonneau - CHU Tours, Tours
  - CH Bretagne Atlantique, Vannes

REFERENCES:
- [Derived] Bourcier R, Marnat G, Dargazanli C, Zhu F, Consoli A, Shotar E, Premat K, Eugene F, Janot K, L'Allinec V, Ognard J, Desilles JP, Blanc R, Gentric JC, Bourdain F, Labreuche J, Liao L, Clarencon F, Barreau X, Ifergan H, Hak JF, Kerleroux B, Pop R, Soize S, Bricout N, Caroff J, Richter JS, Desal H, Lapergue B, Rouchaud A; JENI Research Collaborative. Safety and efficacy of stent retrievers plus contact aspiration in patients with acute ischaemic anterior circulation stroke and positive susceptibility vessel sign in France (VECTOR): a randomised, single-blind trial. Lancet Neurol. 2024 Jul;23(7):700-711. doi: 10.1016/S1474-4422(24)00165-0. PMID 38876748